CLINICAL TRIAL: NCT05301517
Title: A Randomized, Open-label, Active-controlled, Multicenter Phase 3 Study to Investigate the Efficacy and Safety of Roxadustat for Treatment of Anemia in Subjects Receiving Chemotherapy Treatment for Non-Myeloid Malignancies
Brief Title: A Study to Evaluate the Efficacy and Safety of Roxadustat for the Treatment of Anemia in Participants Receiving Chemotherapy Treatment for Non-Myeloid Malignancies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-4592-898
Record Dates: First submitted 2022-03-19; First posted 2022-03-29 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Chemotherapy Induced Anemia
MeSH Terms: interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roxadustat (Experimental): Participants will receive roxadustat, administered orally 3 times per week (TIW) for 12 weeks to achieve Hb levels of 100-120 g/L. The starting dose will be based on the participant's weight group. The maximum dose for individual participants may not exceed 3.5 milligrams (mg)/kilogram (kg) or 400 mg TIW whichever is lower.
  Interventions: Drug: Roxadustat
- SEPO® (Active Comparator): Participants will receive SEPO®, injected subcutaneously TIW for 12 weeks to achieve Hb levels of 100-120 g/L. The starting dose will be 150 international units (IU)/kg subcutaneously TIW.
  Interventions: Drug: SEPO®

INTERVENTIONS:
Drug: SEPO® — SEPO® will be administered per dose and schedule specified in the arm description.
  Other Names: Recombinant human erythropoietin-α [rHuEPO-α]
  Arms: SEPO®
Drug: Roxadustat — Roxadustat will be administered per dose and schedule specified in the arm description.
  Other Names: FG-4592
  Arms: Roxadustat

SUMMARY:
The main goal of this study is to evaluate the efficacy of roxadustat for treatment of anemia in participants with non-myeloid malignancies receiving multi-cycle treatments of myelosuppressive chemotherapy.

DETAILED DESCRIPTION:
Participants who are eligible for participation will be randomized to roxadustat and SEPO® (recombinant human erythropoietin-α [rHuEPO-α]), and undergo a 12-week treatment period followed by a 4-week follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of non-myeloid malignancy, by histological or cytological confirmation.
* Anemia related to myelosuppressive chemotherapy, defined as Hb ≤100 g/L at screening with documented participant's Hb level decrease ≥10 g/L after the initiation of chemotherapy as judged by the investigator.
* Planned concurrent treatment of cancer (myelosuppressive chemotherapy) for at least 8 additional weeks.
* Body weight ≥40 kg.
* Eastern Cooperative Oncology Group (ECOG) performance status of 1 or 2.
* Ferritin ≥50 nanograms (ng)/milliliter (mL) and transferrin saturation (TSAT) ≥10%.

Key Exclusion Criteria:

* Participants with cancer receiving myelosuppressive chemotherapy when the anticipated outcome is cure.
* Participants who are only receiving hormonal products, biological products, novel immunosuppressive products (such as programmed cell death protein-1 [PD-1] and programmed death-ligand 1 [PD-L1] checkpoint inhibitors) or targeted biological or radiation therapy to treat/manage their cancer, however if chemotherapy is co-administered with these products, then it is acceptable to enroll the participant.
* Participants with hematocrit (HCT) ≥36%.
* Participants who have received an RBC transfusion or ESA within 4 weeks of randomization.
* Thromboembolic event (including but not limited to deep vein thrombosis [DVT], pulmonary embolism, myocardial infarction, stroke, transient ischemic attack [TIA] within previous 6 months of screening.
* Clinically significant anemia due to other etiologies such as iron deficiency, vitamin B12 or folate deficiency, autoimmune anemia, hemolysis, hemorrhage, or hereditary anemia such as sickle cell anemia or thalassemia.
* The Investigator judges that the participant will be unable to fully participate in the study and complete it for any reason, including inability to comply with study procedures and treatment, addiction, or any other relevant medical conditions.

Note: Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin (Hb) Level From Baseline to the Level Averaged Over Weeks 9-13 | Baseline, Weeks 9 through 13
  Hb levels measured from Weeks 9 through 13 will be averaged in order to provide a single measure for comparison to the baseline Hb levels.

SECONDARY OUTCOMES:
Percentage of Participants who Achieve a ≥10 Grams (g)/Liter (L) Increase in Hb From Baseline Through Week 13 | Baseline through Week 13
Percentage of Participants who Require Red Blood Cell (RBC) Transfusion or Hb <60 g/L or with any Hb< 60 g/L From Week 5 Through Week 13 | Week 5 through Week 13
Change From Baseline in Functional Assessment of Cancer Therapy-Anemia (FACT-An) Subscale Score Averaged Over Weeks 9-13 | Baseline, Weeks 9 through 13
  FACT-An subscale scores will be averaged over Weeks 9 through 13 in order to provide a single measure for comparison to the baseline score.
Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Subscale Score Averaged Over Weeks 9-13 | Baseline, Weeks 9 through 13
  FACIT-F subscale scores will be averaged over Weeks 9 through 13 in order to provide a single measure for comparison to the baseline score.
Percentage of Participants who Require Dose Reduction or a Dose-Hold of Chemotherapy Due to Anemia | Baseline through Week 13
Change in Hb From Baseline up to 4 Weeks After the Last Dose of Chemotherapy During the Treatment Period | Baseline up to 4 weeks after the last dose of chemotherapy (up to Week 16)
Change in Hb From Baseline Through Week 9 | Baseline through Week 9
Change in Hb From Baseline Through Week 13 | Baseline through Week 13
Percentage of Participants who Achieve a ≥ 15 g/L Increase in Hb From Baseline Through Week 13 | Baseline through Week 13
Percentage of Participants who Achieve Hb Levels ≥ 110 g/L From Baseline Through Week 13 | Baseline through Week 13
Percentage of Participants who Achieve an Increase in Hb of 15 g/L or Attaining a Hb of 110 g/L From Baseline Through Week 13 | Baseline through Week 13
Time to First RBC Transfusion | Baseline up to Week 13
Percentage of Participants Requiring 1 or More RBC Transfusion | Baseline up to Week 13
Number of RBC Transfusions Adjusted for Exposure From Baseline Through Week 13 | Baseline through Week 13
Percentage of Participants who Require RBC Transfusion as Medical Intervention and/or Erythropoiesis-Stimulating Agent (ESA) as a Rescue Agent | Baseline through Week 13

CONTACTS AND LOCATIONS:
Locations (45):
- China (45):
  - Affiliated Hospital of Hebei University, Baoding
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Capital Medical University Chest Hospital, Beijing
  - Peking University Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - Chongqing Bishan People's Hospital, Chongqing
  - The Second Affiliated Hospital of Third Military Medical University (Xinqiao Hospital), Chongqing
  - Deyang People's Hospital, Deyang
  - The First People's Hospital of Foshan, Foshan
  - Fujian Medical University Union Hospital, Fuzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University - Gynecologic Oncology Department, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University - Oncology Department, Guangzhou
  - Hangzhou Cancer Hospital, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Cancer Hospital, Hefei
  - Jiangxi Cancer Hospital, Jiangxi
  - Shandong First Medical University Cancer Hospital, Jinan
  - The Second Hospital of Lanzhou University, Lanzhou
  - Jiangsu Province Hospital, Nanjing
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Neijiang Second People's Hospital, Neijiang
  - Ningbo First Hospital, Ningbo
  - Jiangxi Pingxiang People's Hospital, Pingxiang
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Shanghai Fifth People's Hospital, Shanghai
  - Liaoning Cancer Hospital & Institute, Shenyang
  - The First Hospital of China Medical University - Oncology Department Breast Cancer Group, Shenyang
  - The First Hospital of China Medical University - Oncology Department Lung Cancer Group, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - Shanxi Cancer Hospital, Taiyuan
  - Union Hospital Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - University of Science and Technology, Wuhan
  - Wuhan Fourth Hospital, Wuhan
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Cancer Hospital of Xinjiang Medical University, Xinjiang
  - Xuzhou Central Hospital, Xuzhou
  - Yantai Yuhuangding Hospital, Yantai
  - General Hospital of Ningxia Medical University, Yinchuan
  - Henan Cancer Hospital, Zhengzhou
  - Zhuzhou Central Hospital, Zhuzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu S, Wu J, Jiang J, Guo Q, Yu Y, Liu Y, Zhang H, Qian L, Dai X, Xie Y, Fu T, Lee T, Lu Y, Ma R, Eisner MD. Efficacy and Safety of Roxadustat for Anemia in Patients Receiving Chemotherapy for Nonmyeloid Malignancies: A Randomized, Open-Label, Active-Controlled Phase III Study. J Clin Oncol. 2025 Jan 10;43(2):143-153. doi: 10.1200/JCO.23.02742. Epub 2024 Oct 1. PMID 39353163
- [Derived] Glaspy J, Gabrail NY, Locantore-Ford P, Lee T, Modelska K, Samal V, Henry DH. Open-label, Phase 2 study of roxadustat for the treatment of anemia in patients receiving chemotherapy for non-myeloid malignancies. Am J Hematol. 2023 May;98(5):703-711. doi: 10.1002/ajh.26865. Epub 2023 Feb 24. PMID 36710399